CLINICAL TRIAL: NCT02818829
Title: Biological and Clinical Database for Pancreatic Adenocarcinoma
Acronym: BACAP
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 13 038 07
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Adenocarcinoma; Endoscopic ultrasonography; Fine-needle aspiration; Biomarkers; Epidemiology; DNA tumors
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, saliva, DNA and RNA from tumor cells, tissue from tumor biopsie, tissue from tumor and adjacent tissue of pancreas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Collection of biological samples
  Interventions: Other: Collection of biological samples

INTERVENTIONS:
Other: Collection of biological samples — Collection of biological samples including whole blood, serum, plasma, saliva, DNA and RNA from tumor cells, tissue from tumor biopsies, tissue from tumor and adjacent tissue of pancreas

SUMMARY:
BACAP is a biobank dedicated to the pancreatic adenocarcinoma funded by institut national institue du cancer (INCa) and coordinated by Dr Barbara Bournet from Toulouse hospital. This base includes clinical data and biological samples such as blood, serum, plasma, saliva, DNA and RNA from tumors cells.

The mission of this prospective project is to make available to the scientific community a clinical biological base from patients with pancreatic adenocarcinoma

DETAILED DESCRIPTION:
Pancreatic cancer represents the fifth cause of death by cancer in Western countries. In over 90% of cases, it is due to an adenocarcinoma. The only curative treatment for pancreatic cancer remains the surgical exeresis. This one can only be suggested as a curative treatment in only 10 to 15% of cases. Besides, prevention or screening is impossible due to the absence of clearly identified risk factors or groups and to the absence of useful markers for the diagnosis in clinical practice.

The research efforts in this area must face a double challenge: saving time while improving the diagnosis period and strengthen the therapeutic equipment. It is important to identify and characterise the new molecular markers applicable for a better diagnosis and/or treatment (especially the response factors to chemotherapy). The present project aims at creating a multicentre national network used to set up a clinical biological base (CBB) dedicated to the pancreatic adenocarcinoma, built on the best quality standards, for the biological resources as well as the associated clinical and epidemiological data.

The originality of this CBB relies on the fact that it will have not only tumour tissues sampled from surgical specimens of resectable tumours but also cell and biopsy material from unresectable and/or metastatic tumours sampled under endoscopic ultrasonography (1500 biopsies over 3 years coupled to systematic blood samples). Endoscopic ultrasonography is a technique used to specifically perform biopsies on pancreatic tumours and to obtain useful cell material for research. To these samples will be associated every clinical and epidemiological target data required for research projects related to this unique CBB in France. From these samples, DNA and RNA will be especially isolated, as it is a precious biological material for the programmed molecular analyses.

There are many stakes: creating a French network in order to form, with the prospective plans over 3 years, a collection of tissue, biopsies, nucleic acids from pancreatic cancer associated to circulating blood samples and relevant clinical data. Thanks to this collection, the investigator team hope to be able to identify new molecular markers (from cancer tissue and/or circulating blood from pancreatic cancer patients) applicable to clinical practice to diagnose, to assess the prognosis or to predict the response to pancreatic cancer chemotherapy. The investigator team will also try to identify new risk factors for this cancer, especially regarding the diet. The base will thus be made up from 12 different French centres from University Hospital and private Centres where gastroenterologists, oncologists, digestive surgeons, anatomopathologists, epidemiologists intervene as they are all associated to scientific teams dedicated to pancreatic cancer, itself already formed in collaborative networks.

Investigators hope through this project: to get a unique and exceptional CBB for pancreatic cancer, to reach the required standards (especially Inca) for this CBB, and to be internationally recognised. This base will be a strong guarantee to identify new molecular markers for the diagnosis, the prognosis, and the predictive response to chemotherapy for pancreatic cancer, especially when locally advanced. Finally, the epidemiological projects related to this project are originally about the nutritional issues (regardless of the lipid diet and the cachexia) associated to pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient eighteen years old
* Histologically or cytologically confirmed pancreatic adenocarcinoma
* Solid pancreatic mass explored with tomodensitometry or endoscopic ultrasonography fine-needle aspiration
* Informed consent signed

Exclusion Criteria:

* no informed consent
* pregnancy women
* no histologically or cytologically confirmed pancreatic adenocarcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a pancreatic adenocarcinoma proven cytologically or histologically without any treatment
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Constitution of a transdisciplinary biobank with collection of biological samples with DNA | Through the study completion, an average of 11 months
  The present project aims at creating, coordinating, animating a transdisciplinary multicentric national network, used to set up a clinical biological base (CBB) dedicated to the pancreatic adenocarcinoma
Constitution of a transdisciplinary biobank with collection of biological samples without DNA | Through the study completion, an average of 11 months
  The present project aims at creating, coordinating, animating a transdisciplinary multicentric national network, used to set up a clinical biological base (CBB) dedicated to the pancreatic adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Barbara BOURNET, MD; PHD, Principal Investigator — University Hospital, Toulouse
Locations (16):
- France (16):
  - University Hospital Bordeaux, Bordeaux
  - Beaujon Hospital, Clichy
  - University Hospital Lille, Lille
  - University Hospital of Lille, Lille
  - Centre Léon Bérard, Lyon
  - Private Hospital Jean Mermoz, Lyon
  - Hopital La Timone, Marseille
  - Hospital Nord, Marseille
  - Institut Regional du Cancer de Montpellier, Montpellier
  - University Hospital Montpellier, Montpellier
  - University Hospital of NICE, Nice
  - Saint-Louis Hospital, Paris
  - Clinique du Trocadero, Paris
  - Pau Hospital, Pau
  - University Hospital Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maulat C, Canivet C, Touraine C, Gourgou S, Napoleon B, Palazzo L, Flori N, Piessen G, Guibert P, Truant S, Assenat E, Buscail L, Bournet B, Muscari F, The Bacap Consortium. A New Score to Predict the Resectability of Pancreatic Adenocarcinoma: The BACAP Score. Cancers (Basel). 2020 Mar 25;12(4):783. doi: 10.3390/cancers12040783. PMID 32218346
- [Derived] Frere C, Bournet B, Gourgou S, Fraisse J, Canivet C, Connors JM, Buscail L, Farge D; BACAP Consortium. Incidence of Venous Thromboembolism in Patients With Newly Diagnosed Pancreatic Cancer and Factors Associated With Outcomes. Gastroenterology. 2020 Apr;158(5):1346-1358.e4. doi: 10.1053/j.gastro.2019.12.009. Epub 2019 Dec 14. PMID 31843588
- [Derived] Canivet C, Gourgou-Bourgade S, Napoleon B, Palazzo L, Flori N, Guibert P, Piessen G, Farges-Bancel D, Seitz JF, Assenat E, Vendrely V, Truant S, Vanbiervliet G, Berthelemy P, Garcia S, Gomez-Brouchet A, Buscail L, Bournet B; BACAP Consortium. A prospective clinical and biological database for pancreatic adenocarcinoma: the BACAP cohort. BMC Cancer. 2018 Oct 16;18(1):986. doi: 10.1186/s12885-018-4906-4. PMID 30326968